CLINICAL TRIAL: NCT02967458
Title: Detection of High Grade Prostate Cancer With Subharmonic Ultrasound Imaging, A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor - Radiology, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15F.607; R21CA202214 (NIH); JT 8299 (Other: JeffTrial Number)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prostatic Neoplasm
Keywords: prostate cancer; prostate ultrasound; subharmonic imaging; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate Biopsy Patients (Experimental): Fifty patients who are scheduled for a clinically indicated prostate biopsy, and who are able to undergo contrast enhanced transrectal ultrasound will be included in this single arm study. Each of the study subjects will receive in intravenous infusion of a microbubble contrast agent known as Definity™, (Perflutren Lipid Microsphere, Lantheus Medical Imaging, Inc; N. Billerica, MA). Based upon our previous experience, two vials of Perflutren Lipid Microsphere will be mixed and diluted in 50 ml of normal saline, yielding a concentration of 49.4 μl/ml. For the purpose of contrast-enhanced imaging, Perflutren Lipid Microsphere will be infused over approximately 10-12 minutes, during which time ultrasound imaging and biopsy will be performed.
  Interventions: Drug: Perflutren Lipid Microsphere Intravenous Suspension

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere Intravenous Suspension — The intravenous administration of Perflutren Lipid Microsphere will provide enhancement of vascular tissue when performing subharmonic prostate ultrasound imaging. This enhancement will be used to guide targeted biopsy of the prostate to vascular areas which are more likely to contain aggressive prostate cancer.
  Other Names: Definity™ (Lantheus Medical Imaging, Inc; N. Billerica, MA)

SUMMARY:
This is a phase II single center study using contrast-enhanced ultrasound to identify aggressive forms of prostate cancer with subharmonic imaging.

The following are the study objectives:

1. To implement subharmonic imaging technology on a transrectal probe suitable for prostate imaging and biopsy
2. To demonstrate visualization of prostatic vascularity using subharmonic contrast-enhanced imaging.
3. To provide a preliminary estimate of the diagnostic accuracy of contrast-enhanced subharmonic imaging for detection of clinically significant PCa.

The study will include 50 subjects who are scheduled for prostate biopsy. Each subject will receive an intravenous infusion of microbubble contrast material immediately prior to a prostate biopsy procedure. The study will demonstrate whether subharmonic imaging with a microbubble contrast agent allows for detection of clinically significant prostate cancer.

DETAILED DESCRIPTION:
Background: Prostate cancer (PCa) is the most frequently diagnosed cancer among American males, accounting for 27 % of new cancer diagnoses, but it is directly responsible for only 9.5 % of cancer related deaths. Two recently published clinical trials suggest that overdiagnosis and overtreatment of potentially insignificant cancer is a major drawback of prostate cancer screening, and point to the need for a more specific screening tool that can identify clinically significant prostate cancer. The US-based Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial failed to show a mortality benefit from screening and treatment of prostate cancer. The European Randomized Study of Screening for Prostate Cancer (ERSPC) suggests that with the current standard of care, 1410 men must be screened and 48 additional cases of prostate cancer treated to prevent one death from prostate cancer. Based upon these trials, the U.S. Preventive Services Task Force (USPSTF) has issued a grade "D" recommendation against PSA-based screening for PCa.

Contrast-Enhanced Ultrasound: Recent studies have demonstrated that contrast-enhanced harmonic imaging (HI) can identify enhancement related to vascular flow in higher grade PCa, and that HI can selectively detect patients with "clinically significant" PCa that are most likely to benefit from therapy. Subharmonic imaging (SHI) is a newer technology for contrast-enhanced ultrasound imaging that provides a 10-fold improvement in the signal to background ratio for visualization of small vascular structures, but has not been previously implemented on a transrectal ultrasound probe. SHI of the prostate is expected to advance the imaging of prostatic neovascularity and to improve selective biopsy of clinically significant PCa.

Objective: To adapt SHI to a transrectal probe appropriate for prostate imaging and biopsy (over the first 6 months of this study). The subsequent 18 month pilot clinical study will enroll 50 participants who have a clinical indication for prostate biopsy to quantify SHI for the detection of clinically significant PCa (defined as: Gleason score ≥ 7, a single core with > 50 % involvement, or > 25 % of biopsy cores positive for PCa).

Approach: Each participant will undergo a transrectal ultrasound evaluation of the prostate with conventional grayscale and color Doppler imaging, as well as contrast-enhanced imaging with color Doppler, HI and SHI approaches. Imaging results from each of these techniques will be recorded, but only the SHI findings will be used to guide a targeted biopsy of the prostate. A maximum of 6 targeted biopsy cores will be obtained from each participant, based upon suspicious areas identified with SHI. Following the targeted biopsy, each participant will also receive a 12-part systematic biopsy consisting of 6 laterally directed biopsy cores and 6 medially directed biopsy cores. The pilot study is designed to estimate the detection of clinically significant cancer that will be obtained with targeted biopsy based upon SHI along with the medially directed systematic sextant biopsy cores (≤ 12 cores total).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be scheduled for a clinically indicated needle biopsy of the prostate based upon an elevated PSA, abnormal digital rectal examination, or based upon active surveillance of prostate cancer.
2. Subject must be able and willing to give written informed consent for a contrast enhanced ultrasound study of the prostate.
3. Subject must be a male at least 18 years of age when informed consent is obtained.
4. Subject must have a life expectancy that exceeds the duration of the clinical trial.

Exclusion Criteria:

1. Participant in a clinical trial involving an investigational drug within the past 30 days.
2. Prior allergic reaction to the ultrasound contrast agent Definity™
3. Previous treatment for PCa.
4. Clinically unstable, severely ill, or moribund.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan J Halpern, MD, Principal Investigator — Thomas Jefferson University; Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halpern EJ, Gomella LG, Forsberg F, McCue PA, Trabulsi EJ. Contrast enhanced transrectal ultrasound for the detection of prostate cancer: a randomized, double-blind trial of dutasteride pretreatment. J Urol. 2012 Nov;188(5):1739-45. doi: 10.1016/j.juro.2012.07.021. Epub 2012 Sep 19. PMID 22998915
- [Background] Aigner F, Schafer G, Steiner E, Jaschke W, Horninger W, Herrmann TR, Nagele U, Halpern EJ, Frauscher F. Value of enhanced transrectal ultrasound targeted biopsy for prostate cancer diagnosis: a retrospective data analysis. World J Urol. 2012 Jun;30(3):341-6. doi: 10.1007/s00345-011-0809-6. Epub 2011 Dec 18. PMID 22179312
- [Background] Trabulsi EJ, Sackett D, Gomella LG, Halpern EJ. Enhanced transrectal ultrasound modalities in the diagnosis of prostate cancer. Urology. 2010 Nov;76(5):1025-33. doi: 10.1016/j.urology.2010.05.022. Epub 2010 Aug 16. PMID 20719368
- [Background] Nelson ED, Slotoroff CB, Gomella LG, Halpern EJ. Targeted biopsy of the prostate: the impact of color Doppler imaging and elastography on prostate cancer detection and Gleason score. Urology. 2007 Dec;70(6):1136-40. doi: 10.1016/j.urology.2007.07.067. PMID 18158034
- [Background] Linden RA, Trabulsi EJ, Forsberg F, Gittens PR, Gomella LG, Halpern EJ. Contrast enhanced ultrasound flash replenishment method for directed prostate biopsies. J Urol. 2007 Dec;178(6):2354-8. doi: 10.1016/j.juro.2007.08.022. Epub 2007 Oct 22. PMID 17936814
- [Background] Halpern EJ, Ramey JR, Strup SE, Frauscher F, McCue P, Gomella LG. Detection of prostate carcinoma with contrast-enhanced sonography using intermittent harmonic imaging. Cancer. 2005 Dec 1;104(11):2373-83. doi: 10.1002/cncr.21440. PMID 16240450

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostate Biopsy Patients: Fifty five patients who are scheduled for a clinically indicated prostate biopsy, and who are able to undergo contrast enhanced transrectal ultrasound will be included in this single arm study. Each of the study subjects will receive in intravenous infusion of a microbubble contrast agent known as Definity™, (Perflutren Lipid Microsphere, Lantheus Medical Imaging, Inc; N. Billerica, MA). Based upon our previous experience, two vials of Perflutren Lipid Microsphere will be mixed and diluted in 50 ml of normal saline, yielding a concentration of 49.4 μl/ml. For the purpose of contrast-enhanced imaging, Perflutren Lipid Microsphere will be infused over approximately 10-12 minutes, during which time ultrasound imaging and biopsy will be performed.
Period: Overall Study
Arm/Group | Prostate Biopsy Patients
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prostate Biopsy Patients
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Prostate Cancer Was Detected With Subharmonic Imaging
Description: The initial phase of the trial will develop and test subharmonic imaging to demonstrate enhanced visualization of prostate vascularity in all study participants. We will report the percentage of study subjects in whom visualization of prostate vascularity is increased with subharmonic imaging.
Time Frame: One week from baseline
Measure: Count of Participants; unit: Participants
Groups:
- 1Prostate Biopsy Patients: Patients who are scheduled for a clinically indicated prostate biopsy, and who are able to undergo contrast enhanced transrectal ultrasound will be included in this single arm study. Each of the study subjects will receive in intravenous infusion of a microbubble contrast agent known as Definity™, (Perflutren Lipid Microsphere, Lantheus Medical Imaging, Inc; N. Billerica, MA). Based upon our previous experience, two vials of Perflutren Lipid Microsphere will be mixed and diluted in 50 ml of normal saline, yielding a concentration of 49.4 μl/ml. For the purpose of contrast-enhanced imaging
  Perflutren Lipid Microsphere Intravenous Suspension: The intravenous administration of Perflutren Lipid Microsphere will provide enhancement of vascular tissue when performing subharmonic prostate ultrasound imaging. This enhancement will be used
Arm/Group | 1Prostate Biopsy Patients
Number analyzed (Participants) | 55
Participants | 24

2. Primary Outcome: Percentage of Biopsy Cores in Which Prostate Cancer Was Detected Using Subharmonic Imaging
Description: Study subjects will be scanned with subharmonic imaging during infusion of the microbubble contrast agent. Imaging results will be compared to pathology on prostate biopsy.
Time Frame: One week from baseline
Measure: Number; unit: percentage of biopsy cores
Groups:
- Prostate Biopsy Patients: Patients who are scheduled for a clinically indicated prostate biopsy, and who are able to undergo contrast enhanced transrectal ultrasound will be included in this single arm study. Each of the study subjects will receive in intravenous infusion of a microbubble contrast agent known as Definity™, (Perflutren Lipid Microsphere, Lantheus Medical Imaging, Inc; N. Billerica, MA). Based upon our previous experience, two vials of Perflutren Lipid Microsphere will be mixed and diluted in 50 ml of normal saline, yielding a concentration of 49.4 μl/ml. For the purpose of contrast-enhanced imaging.
  Perflutren Lipid Microsphere Intravenous Suspension: The intravenous administration of Perflutren Lipid Microsphere will provide enhancement of vascular tissue when performing subharmonic prostate ultrasound imaging. This enhancement will be used
Arm/Group | Prostate Biopsy Patients
Number analyzed (Participants) | 55
percentage of biopsy cores | 8.33

3. Primary Outcome: Percentage of Subjects With Previously Unidentified Prostate Cancer Using Magnetic Resonance Imaging
Description: as for outcome 2
Time Frame: One week from baseline
Population: Thirty one subjects of the total 55 had prior negative MRI or negative MRI guided biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Biopsy Patients
Number analyzed (Participants) | 31
Participants | 9

ADVERSE EVENTS:
Time Frame: Assessed for 30 minutes post-injection
Groups:
- Prostate Biopsy Patients: Patients who are scheduled for a clinically indicated prostate biopsy, and who are able to undergo contrast enhanced transrectal ultrasound will be included in this single arm study. Each of the study subjects will receive in intravenous infusion of a microbubble contrast agent known as Definity™, (Perflutren Lipid Microsphere, Lantheus Medical Imaging, Inc; N. Billerica, MA). Based upon our previous experience, two vials of Perflutren Lipid Microsphere will be mixed and diluted in 50 ml of normal saline, yielding a concentration of 49.4 μl/ml. For the purpose of contrast-enhanced imaging, Perflutren Lipid Microsphere will be infused over approximately 10-12 minutes, during which time ultrasound imaging and biopsy will be performed.
  Perflutren Lipid Microsphere Intravenous Suspension: The intravenous administration of Perflutren Lipid Microsphere will provide enhancement of vascular tissue when performing subharmonic prostate ultrasound imaging. This enhancement will be used
Arm/Group | Prostate Biopsy Patients
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 2/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Biopsy Patients (N=55)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Throat Tightness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT02967458/Prot_SAP_000.pdf